CLINICAL TRIAL: NCT03299556
Title: Effect of Wearable Health Technology on Patients Treated for Chronic Pain at Geisinger Health System
Status: Completed | Type: Observational
Sponsor: Purdue Pharma LP (Industry)
Collaborators: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0196
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain
Keywords: Wearable Health Technology; iPhone; Apple Watch; Pain Medication
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- WHT: The WHT group includes only patients newly enrolled in the Geisinger MPP program who consent to participate in the study. WHT subjects will be recruited over 1 year, with 1 year of follow-up.
  Interventions: Other: WHT
- Historic Control: Patients who were enrolled in the MPP in the preceding year. These patients received the MPP educational program but received no WHT as part of their treatment.
- Concurrent Control: Patients being treated for chronic pain in the Geisinger Medical Pain Management (MPM) program over the same time period as the WHT group. These subjects do not receive the MPP educational program nor use WHT as part of their treatment

INTERVENTIONS:
Other: WHT — Incorporating WHT into treatment for chronic pain. WHT includes patient and provider tracking of patient-reported pain, pain management, medication usage, functionality, depression, activity and sleep (measured by 3 axis actigraph); as well as prompts to subjects to engage in self-care, including non-pharmaceutical pain management therapies consistent with MPP training.
  Groups: WHT

SUMMARY:
This is a proof of concept study to measure the effect of Wearable Health Technology (WHT), including the Apple Watch, iPhone, Pain App and Provider Dashboards on important clinical outcomes in patients treated for chronic pain. WHT will be tested in a group of chronic pain patients treated at a specialty pain clinic, the Geisinger Multidisciplinary Pain Program (MPP). Primary and secondary outcomes include pain, physical function, depression, pain medicine use, amount of sleep, activity levels, healthcare resource utilization and cost. The WHT will collect self-reported data on pain, pain management therapies, and medication utilization, and passively collected data on subject activity levels and sleep. Additional data will be collected on device utilization by patients and health care professionals.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, non-blinded trial with historic and concurrent controls to assess the effect of the addition of WHT on patient and health system outcomes. WHT used in this study are the Apple Watch and iPhone, a pain application (Pain App) designed specifically for this study to be used with the watch and phone, and physician and patient dashboards also designed for this study to provide subjects and health care providers data displays of information captured by the WHT.

The WHT will consist of:

* AppleWatch and iPhone
* Patient and provider tracking of patient-reported pain, pain management, medication usage, functionality, depression, activity and sleep (measured by 3 axis actigraph)
* Prompts to subjects to engage in self-care, including non-pharmaceutical pain management therapies consistent with MPP training

Subjects will use the WHT 20 hours per day, every day for a period of 12 months.

Subjects will attend study visits at baseline and months 2, 4, 6, 8, 10 and 12.

Outcome data for control groups will be collected retrospectively from the electronic health record (EHR). Assessments will have occurred as part of their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the MPP
* Completion of the 3-day MPP training
* Ability to understand and complete the informed consent form prior to the initiation of any study procedures
* Adequate motor skills needed to utilize WHT
* Willingness to utilize personal electronic devices and WHT, as expressed and documented during the informed consenting process
* Ability to understand spoken and written English

Exclusion Criteria:

* Cancer diagnosis, AIDS, end-stage liver disease or end-stage renal disease
* Hospitalization >30 days during the 12 months prior to Index Date
* Nursing home or hospice care during the 12 months prior to Index Date
* Presence of an EHR Diagnosis description "OPT-OUT CENTER RESEARCH" which indicates the subject has opted out of (i.e., does not wish to be included in) any Geisinger retrospective research
* Has a terminated Medicine Use Agreement on their Problem List, indicator for substance abuse/dependence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Geisinger chronic pain patients, currently or previously enrolled in the MPP or currently receiving treatment in the MPM program.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Alfieri, PhD, Study Director — Purdue Pharma LP; John J Han, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Long-term Use of Wearable Health Technology by Chronic Pain Patients — https://journals.lww.com/clinicalpain/Fulltext/2022/12000/Long_term_Use_of_Wearable_Health_Technology_by.1.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Wearable Health Tracker (WHT): The WHT group includes only patients newly enrolled in the Geisinger Multidisciplinary Pain Program (MPP) who consent to participate in the study. WHT subjects will be recruited over 1 year, with 1 year of follow-up.
- Historic Control (MPP): Patients who were enrolled in the Multidisciplinary Pain Program (MPP) in the preceding year. These patients received the MPP educational program but received no WHT as part of their treatment.
- Concurrent Control (MPM): Patients being treated for chronic pain in the Geisinger Medical Pain Management (MPM) program over the same time period as the WHT group. These subjects do not receive the MPP educational program nor use WHT as part of their treatment.
Period: Overall Study
Arm/Group | Wearable Health Tracker (WHT) | Historic Control (MPP) | Concurrent Control (MPM)
Started | 113 | 146 | 161
Completed | 105 | 146 | 161
Not Completed | 8 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wearable Health Tracker (WHT) | Historic Control (MPP) | Concurrent Control (MPM) | Total
Number analyzed (Participants) | 105 | 146 | 161 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (12.8) | 50.4 (11.8) | 47.1 (12.5) | 49.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 93 | 110 | 284
  Male | 24 | 53 | 51 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 8 | 15
  Not Hispanic or Latino | 102 | 142 | 153 | 397
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 9 | 17
  White | 102 | 139 | 151 | 392
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Numerical Pain Score (NPS)
Description: self reported 11-point pain scale. The numeric pain score (NPS) is self-reported by the patient on a scale of 0 to 10, with the following scale labels: no pain (0), mild pain (2), moderate pain (4), severe pain (6), very severe pain (8), and worst pain possible (10).
Time Frame: Baseline, 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wearable Health Tracker (WHT) | Historic Control (MPP) | Concurrent Control (MPM)
Number analyzed (Participants) | 79 | 135 | 139
score on a scale
  Baseline | 5.48 (1.50) | 6.50 (1.57) | 6.48 (1.70)
  12-month follow-up | 5.22 (1.53) | 6.10 (1.36) | 6.15 (1.54)

2. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: self reported measurement of depression. The scale ranges from 0 to 27, indicating the following levels of depression severity: none (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27).
Time Frame: Baseline, 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wearable Health Tracker (WHT) | Historic Control (MPP) | Concurrent Control (MPM)
Number analyzed (Participants) | 33 | 75 | 31
score on a scale
  Baseline | 14.07 (5.65) | 15.19 (6.34) | 14.63 (4.90)
  12-month follow-up | 11.78 (6.18) | 12.89 (6.25) | 11.31 (5.73)

3. Primary Outcome: Mean Daily Morphine Equivalents (MEQs)
Description: calculated from health records, average amount of daily pain medication [as measured by the daily milligrams of morphine equivalents (MME)].
Time Frame: Baseline, 12-month follow-up
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Wearable Health Tracker (WHT) | Historic Control (MPP) | Concurrent Control (MPM)
Number analyzed (Participants) | 39 | 74 | 84
MME
  Baseline | 51.38 (44.84) | 56.83 (76.30) | 43.42 (68.62)
  12-month follow-up | 38.36 (34.88) | 54.46 (66.51) | 43.69 (51.39)

4. Secondary Outcome: Oswestry Disability Index (ODI)
Description: self reported measure of functionality, related to back and neck pain. The ODI is a self-administered questionnaire assessing symptoms and severity of back or neck pain on a scale from 0 to 100. This measurement evaluates the loss of function in activities of daily living. Two ODI questionnaires were used in this study, one for neck pain and one for back pain. Interpretation of ODI scoring is as follows: minimal disability (0-20), moderate disability (21-40), severe disability (41-60), and crippled (61-80). Scores over 80 suggest the patient may be bedbound or exaggerating their symptoms and careful evaluation is recommended.
Time Frame: Baseline, 12-month follow-up
Population: The numbers analyzed differ because two different measures were used - the ODI Back was administered only to patients with back pain, the ODI Neck was administered only to patients with neck pain.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wearable Health Tracker (WHT) | Historic Control (MPP) | Concurrent Control (MPM)
Number analyzed (Participants) | 54 | 80 | 36
score on a scale
  ODI (Back) Baseline | 47.67 (13.54) | 55.05 (12.43) | 51.20 (11.78)
  ODI (Back) 12-month follow-up | 45.46 (14.38) | 53.99 (12.99) | 46.28 (16.74)
  ODI (Neck) Baseline: number analyzed (Participants) | 35 | 58 | 27
  ODI (Neck) Baseline | 50.07 (14.51) | 59.23 (13.96) | 53.10 (13.70)
  ODI (Neck) 12-month follow-up: number analyzed (Participants) | 35 | 58 | 27
  ODI (Neck) 12-month follow-up | 51.03 (14.50) | 59.59 (13.79) | 51.40 (17.27)

5. Other Pre Specified Outcome: Activity Levels (WHT Group Only)
Description: number of daily steps as measured by WHT application. Insufficient data collected for analysis of this outcome measure.
Time Frame: 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Sleep (WHT Group Only)
Description: quantity (hours) and quality as measured by WHT application. Insufficient data collected for analysis of this outcome measure.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 12 months for participants in the WHT group. Up to a 12-month retrospective review of AE data was performed for the patients in the MPP and MPM control groups.
Arm/Group | Wearable Health Tracker (WHT) | Historic Control (MPP) | Concurrent Control (MPM)
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/146 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/146 | 0/161
Other Adverse Events (participants affected / at risk) | 0/113 | 0/146 | 0/161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT03299556/Prot_SAP_000.pdf